CLINICAL TRIAL: NCT03795363
Title: Nutritional Impact of Orkambi Treatment in 2 to 5 Year Old Children Homozygous for F508del Mutations
Brief Title: Orkambi Treatment in 2 to 5 Year Old Children With CF
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-015669
Record Dates: First submitted 2018-12-28; First posted 2019-01-07 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Cystic Fibrosis
Keywords: CF; CFTR; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Orkambi — Orkambi is a novel approved therapy for use in people homozygous for the F508del mutation in the CFTR gene. It is a combination of lumacaftor (VX-809) and ivacaftor( VX-770) that addresses both the processing and gating defects of the F508del mutation. The small-molecule corrector lumacaftor corrects the F508del processing defect and increases epithelial delivery of CFTR protein1. Ivacaftor is a CFTR potentiator that increases the channel open probability in F508del-mutant CFTRs that undergo epithelial delivery in vitro and has an additive effect with lumacaftor on chloride transport (2,3,4,5).

SUMMARY:
The purpose of this observational research study is to determine the effects of clinically prescribed Orkambi treatment on 2 to 5 year old children homozygous for the F508del Mutations in the Cystic fibrosis transmembrane conductance regulator (CFTR) gene on sleeping energy expenditure, growth status and gut health and function.

DETAILED DESCRIPTION:
Orkambi is a novel FDA approved (August, 2018) therapy for use in patients with cystic fibrosis (CF) who are 2 to 5 years of age and homozygous for F508del mutations in the CFTR gene. It is a combination of lumacaftor and ivacaftor that addresses both the processing and gating defects of the F508del mutation. This investigator-initiated study is designed to evaluate the nutritional, growth and GI impact of Orkambi treatment for this unique younger (2 to 5 years) patient cohort. This proposal extends previous highly informative nutrition and weight gain investigation of ivacaftor treatment in people with CF gating mutations to another CFTR modulator treatment (Orkambi) in people homozygous for F508del mutations. The primary aims of the study are to evaluate the impact of 24 weeks of Orkambi treatment in 2 to 5 year old subjects with CF homozygous for F508del mutations on sleeping or resting energy expenditure, growth status and gut health and function in n=32 children ages 2.0 to 5.9 years of age. Protocol evaluations will occur at baseline (pre-treatment) and 12 and 24 weeks after clinically prescribed Orkambi treatment has begun. Other outcomes of significant clinical interest in young subjects with CF will be explored. All subjects will be evaluated as outpatient at The Children's Hospital of Philadelphia, and will be recruited both regionally and nationally to ensure timely enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis and homozygous for F508del mutations, approved for treatment
* Age: 2.0 to 5.9 years
* In usual state of good health
* A clinical decision has been made for subject to begin Orkambi treatment
* Family committed to the 6 to 8 month study protocol with visits to the Children's Hospital of Philadelphia (CHOP) that will last 2-3 days for the baseline visit (Visit 1) prior to Orkambi and the 24 week visit (Visit 3) after clinically prescribed Orkambi treatment has begun, and will last up to 2 days for the 12 week visit (Visit 2) after Orkambi treatment has begun.

Exclusion Criteria:

* On parenteral nutrition
* Use of any medications that inhibit or induce cytochrome P450 (CYP) 3A
* Liver function tests elevated above 3x the reference range for age and sex
* Lung disease considered severe based on clinical impression by home CF center.
* Other illness affecting growth or nutritional status
* Other contraindications described for Orkambi therapy

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 2 to 5 year old subjects with a diagnosis of cystic fibrosis and homozygous for F508del mutations and who are in a usual state of good health with a clinical decision to start orkambi treatment.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Sleeping or Resting Energy Expenditure | 24 Weeks
  Investigators will examine the effects of 24 weeks of orkambi treatment on subject's SEE (sleeping energy expenditure) or REE (resting energy expenditure). Using indirect calorimetry, SEE/REE will be assessed using a computerized metabolic cart Vmax ENCORE at each protocol visit while the child is asleep or resting quietly. SEE/REE will be assessed in the morning if possible and careful note of previous feeding of the child, including the time of day, amount of food, and feeding interval prior to test. It will depend on the age of the subject, and if the subject still takes daily naps and is able to rest quietly without moving, if they will perform sleeping energy expenditure or resting energy expenditure. This will be one outcome measure for each subject, and it will depend on if the subject can nap (SEE) or rest quietly without moving (REE).
Anthropometric Assessment | 24 Weeks
  Investigators will examine the effects of 24 weeks of orkambi treatment on subject's body mass index (BMI). Investigators will compare the results to BMI Z scores over 24 weeks compared to baseline.

SECONDARY OUTCOMES:
Fecal Elastase I/Pancreatic Function | 24 Weeks
  Investigators will examine the effects of 24 weeks of orkambi treatment on subject's pancreatic function. Pancreatic function will be assessed at two visits by obtaining spot stool samples with fecal elastase 1. The concentration of fecal elastase I is indicative of pancreatic function.
Fecal Calprotectin/Gut Inflammation | 24 Weeks
  Investigators will examine the effects of 24 weeks of orkambi treatment on subject's fecal calprotectin concentration. Spot stool samples will be obtained to determine fecal calprotectin concentration, which is a marker for gut inflammation.
Plasma Total Fatty Acids | 24 Weeks
  Investigators will examine the effects of 24 weeks of orkambi treatment on subject's dietary fat absorption. A total plasma fatty acid panel will be assessed to measure the change in status of 22 fatty acids.

OTHER OUTCOMES:
Dietary Intake | 24 Weeks
  Three day weighed food record will be obtained and to determine changes in dietary caloric intake and micro and macronutrient intake over the course of 24 weeks on orkambi treatment.
Serum fat soluble vitamin levels | 24 Weeks
  Investigators will examine the changes in serum fat soluble vitamin A, E, D and K concentration levels after 24 weeks of orkambi treatment.
Changes in bile acid concentration levels | 24 Weeks
  Investigators will examine changes in the concentration levels of 14 bile acid species in subjects over the course of 24 weeks on orkambi treatment.
Changes in concentration levels of serum calprotectin | 24 Weeks
  Investigators will examine changes in the concentration levels of serum calprotectin in subjects over the course of 24 weeks on orkambi treatment.
Muscle-Fat Stores | 24 Weeks
  Investigators will measure body composition to determine muscle and fat store changes over the course of 24 weeks on orkambi treatment compared to baseline.
Growth status changes | 24 Weeks
  Investigators will observe the changes in growth status over time. Growth status will be measured by determining the changes in three different measurements- length (cm), weight (kg) and head circumference (cm). Each value will be used to calculate BMI (kg/cm^2), which will be used in accordance with age to determine the growth velocity percentile of the subjects over the course of 24 weeks on orkambi treatment. The growth velocity percentile will be indicative of changes in growth status over time.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Stallings, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Stallings VA, Sainath N, Oberle M, Bertolaso C, Schall JI. Energy Balance and Mechanisms of Weight Gain with Ivacaftor Treatment of Cystic Fibrosis Gating Mutations. J Pediatr. 2018 Oct;201:229-237.e4. doi: 10.1016/j.jpeds.2018.05.018. Epub 2018 Jul 18. PMID 30029855
- [Background] Flume PA, Liou TG, Borowitz DS, Li H, Yen K, Ordonez CL, Geller DE; VX 08-770-104 Study Group. Ivacaftor in subjects with cystic fibrosis who are homozygous for the F508del-CFTR mutation. Chest. 2012 Sep;142(3):718-724. doi: 10.1378/chest.11-2672. PMID 22383668
- [Background] Van Goor F, Hadida S, Grootenhuis PD, Burton B, Cao D, Neuberger T, Turnbull A, Singh A, Joubran J, Hazlewood A, Zhou J, McCartney J, Arumugam V, Decker C, Yang J, Young C, Olson ER, Wine JJ, Frizzell RA, Ashlock M, Negulescu P. Rescue of CF airway epithelial cell function in vitro by a CFTR potentiator, VX-770. Proc Natl Acad Sci U S A. 2009 Nov 3;106(44):18825-30. doi: 10.1073/pnas.0904709106. Epub 2009 Oct 21. PMID 19846789
- [Background] Milla CE, Ratjen F, Marigowda G, Liu F, Waltz D, Rosenfeld M; VX13-809-011 Part B Investigator Group *. Lumacaftor/Ivacaftor in Patients Aged 6-11 Years with Cystic Fibrosis and Homozygous for F508del-CFTR. Am J Respir Crit Care Med. 2017 Apr 1;195(7):912-920. doi: 10.1164/rccm.201608-1754OC. PMID 27805836
- [Background] Wainwright CE, Elborn JS, Ramsey BW. Lumacaftor-Ivacaftor in Patients with Cystic Fibrosis Homozygous for Phe508del CFTR. N Engl J Med. 2015 Oct 29;373(18):1783-4. doi: 10.1056/NEJMc1510466. No abstract available. PMID 26510034
- [Background] Energy and protein requirements. Report of a joint FAO/WHO/UNU Expert Consultation. World Health Organ Tech Rep Ser. 1985;724:1-206. No abstract available. PMID 3937340
- [Background] Schofield WN. Predicting basal metabolic rate, new standards and review of previous work. Hum Nutr Clin Nutr. 1985;39 Suppl 1:5-41. PMID 4044297
- [Background] World Health Organization. WHO Child Growth Standards: Length/height-for-age, weight-for-age, weight-for-length, weight-for-height, and body mass index-for-age. Geneva, Switzerland: WHO Press, World Health Organization; 2006.
- [Background] Borowitz D, Baker SS, Duffy L, Baker RD, Fitzpatrick L, Gyamfi J, Jarembek K. Use of fecal elastase-1 to classify pancreatic status in patients with cystic fibrosis. J Pediatr. 2004 Sep;145(3):322-6. doi: 10.1016/j.jpeds.2004.04.049. PMID 15343184
- [Background] Borowitz D, Lin R, Baker SS. Comparison of monoclonal and polyclonal ELISAs for fecal elastase in patients with cystic fibrosis and pancreatic insufficiency. J Pediatr Gastroenterol Nutr. 2007 Feb;44(2):219-23. doi: 10.1097/MPG.0b013e31802c41de. PMID 17255835
- [Background] O'Connor MG, Seegmiller A. The effects of ivacaftor on CF fatty acid metabolism: An analysis from the GOAL study. J Cyst Fibros. 2017 Jan;16(1):132-138. doi: 10.1016/j.jcf.2016.07.006. Epub 2016 Jul 26. PMID 27473897
- [Background] World Health Organization. WHO Child Growth Standards: Head circumference-for-age, arm circumference-for-age, triceps skinfold-for-age, and subscapular skinfold-for-age. Geneva, Switzerland: WHO Press, World Health Organization; 2007.
- [Background] WHO Multicenter Growth Reference Study Group. WHO Child Growth Standards: Growth Velocity Based on Weight, Length and Head Circumference: Methods and Development. Geneva, Switzerland: WHO Press: World Health Organization; 2009.

DOCUMENTS (2):
  • Study Protocol (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT03795363/Prot_000.pdf
  • Informed Consent Form (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT03795363/ICF_001.pdf